CLINICAL TRIAL: NCT05823649
Title: Effect of Early Versus Delayed Postoperative Feeding in Lower Limb Fracture Surgery: a Randomized Controlled Trial
Brief Title: Effect of Early Versus Delayed Postoperative Feeding in Lower Limb Fracture Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Armed Police Force Hospital, Nepal (Other Government)
Collaborators: Nepal Orthopedic Hospital, Kathmandu, Nepal (Unknown)
Responsible Party: Principal Investigator, Dev Ram Sunuwar, Dietitian and Researcher, Armed Police Force Hospital, Nepal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Postoperative feeding
Record Dates: First submitted 2023-03-20; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Lower Limb Fracture
Keywords: Postoperative diet; Early feeding; Delayed feeding; Lower limb fracture

STUDY DESIGN:
Intervention Model Description: Oral feeding
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early feeding/intervention group (Experimental): The postoperative patients will be intervened after one to two hours from the entry of the patients to the postoperative ward.
  Interventions: Dietary Supplement: Early feeding/intervention group
- Delayed feeding/control group (Active Comparator): The postoperative patients will be fed delayed as traditionally practiced for long time as per the hospital's protocol that breaks the postoperative fasting only after four to six hours of the surgery according to the patient condition. The guideline of the hospital recommends the patients to drink black tea as first postoperative feeding and then facilitated by the semi-solid diet, especially mushy rice which is generally cooked by mixture of rice, vegetables and pulses with salt and a lot of water.
  Interventions: Dietary Supplement: Early feeding/intervention group

INTERVENTIONS:
Dietary Supplement: Early feeding/intervention group — The patients will be given orally 5 to 10 ml of warm water as first feeding. If there will be no problem of swallowing and other clinical complication, they will be further provided 20 ml of water after 10 minutes. If further patients do not suffer from nausea, vomiting and other discomfort, 100 ml clear fluid or less than it will be provided as based on the protocol followed by the study. We will use oral rehydration solution (ORS) as clear fluid.

SUMMARY:
The treatment of lower limb fracture accounting one third of total fracture is a complex problem for the surgical and rehabilitation team. Patients are kept in long term fasting after surgery to prevent from postoperative complications, but it leads to the surgical catabolism resulting delaying the desired improvement in patients. To our knowledge, it has not been widely implemented in clinical settings. Therefore, the aim of the study is to evaluate the effect of early versus delayed postoperative oral feeding in lower limb fracture surgery under regional block anesthesia.

This study utilize single-center, hospital based, open-label, parallel group randomized controlled trial to assess the effect of early postoperative oral feeding in two hours after the surgery over the conventionally delayed feeding. A representative sample size of 275 patients (control group=138 and study group =137) aged 18 years and above having lower limb fracture operated under regional block will be selected for research. The pre-operative nutritional status will be identified with Simplified Nutritional Appetite Questionnaire (SNAQ) and the post-operative outcomes will be measured by Numerical Rating Scale (NRS) system. Preoperative as well as postoperative hand grip strength and Neutrophil Lymphocyte Ratio (NLR) will be assessed. Statistical analysis will be performed using chi square test, Student two sample t-test to compare between the outcome of study and control groups. The outcome of the study may provide an empirical evidence to the anesthesiologists and surgeons towards the emerging concept of postoperative early oral feeding practice in lower limb fracture surgery in clinical settings.

DETAILED DESCRIPTION:
Orthopedic conditions are the physical injuries related to the musculoskeletal system of an individual. The overall incidence of musculoskeletal injury in low- and lower-middle income countries (LMICs) range from 779 to 1574 per 100,000 person-years. Fracture is one of the main cause of injury showing 1,229 per 100,000 individuals. The most common injury due to the road traffic accident was the 69 % fracture with fractures of tibia/fibula accounted as 30.3%. The road traffic injury (RTI) in Nepal for the period 2001-2013 also revealed that the most common fractures are lower extremities and upper extremities. About one third of the total fracture accounted for lower limb fracture and its complications lead to reason for hospital stay. Surgical management for the lower extremities fracture allows quick stabilization of fractures and early mobilization, hence accelerates the return to usual daily life activities. In fact, lower extremities fracture is a complex problem for the surgical and rehabilitation team. Pain as postoperative outcome is associated with many factors like age, duration of surgery, type of surgery, site of surgery, use of anesthesia, ethnicity, and others. Nutritional status is a strong predictor of postoperative outcomes in orthopedics for the preservation of muscle mass, strength and functionality of movement, and therefore it is recognized as an important component of surgical recovery programs. Nutritional assessment includes subjective as well as objective parameters. There are many tools for examining malnutrition and nutritional assessment as subjective parameters. Similarly, different laboratory markers such as albumin, pre-albumin, total lymphocytes, total cholesterol, C-reactive protein, transferrin are considered the objective parameter for the nutritional status evaluation. Higher the pre- and postoperative Neutrophil Lymphocyte Ratio (NLR) is associated with a higher long-term mortality risk in hip fracture surgery in elder people. Nutritional intervention is crucial for enhanced recovery after surgery. Preoperative carbohydrate loading as nutritional intervention is one component of Enhanced Recovery after Surgery (ERAS) which reduces insulin resistivity and postoperative infection. Another study found that preoperative carbohydrate loading in femur fracture has facilitated the ambulatory function, reduced the postoperative pain and hence reduced the length of hospital stay.

Patients are kept in long term fasting after surgery to prevent from postoperative complications. In fact, postoperative fasting leads to surgical catabolism and has increased the ICU stay among cancer patients undergoing elective cancer surgery. Early feeding after surgery challenges the concept of increased incidence of nausea and vomiting, and so late re-feeding has no advantages. Immediate postoperative re-feeding in orthopedic surgery is safe. Earlier post-operative feeding reduce the infection complications, improve healing, and decrease length of stay, so oral feeding should be resumed as soon as possible after surgery, with the goal of returning to solid foods within 24 hours. Previous study found that around 25 gram of essential amino acid can be fed orally within 30 minutes after surgery to facilitate the injury recovery and rehabilitation among athletes. A randomized controlled trial shows that early postoperative feeding at 4 hours is safe, and the traditional policy of starting feeding after 8 hours is outmoded under general anesthesia in orthopedics. The recommendation 5 of European Society for Clinical Nutrition and Metabolism (ESPEN) which states that enteral feeding can be initiated immediately after surgery. However, postoperative patients are mostly re-fed only after 4-6 hours of the surgery followed by the regional anesthesia (spinal, epidural or nerve block). Therefore, the study is intended to evaluate the effect of early postoperative oral feeding in the lower limb fracture surgery under regional block anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 60 years undergoing the lower limb fracture surgery under regional anesthesia
* Intermediate to major categories of surgeries
* American Society of Anesthesiologists (ASA) I and II

Exclusion Criteria:

* Cognitive dysfunction
* Pathological fracture
* Fracture more than one site
* Redo/follow-up surgery
* Unanticipated intraoperative complications
* Use of intraoperative drugs that causes the postoperative nausea and vomiting
* Gastrointestinal disorder such as peptic ulcer, hiatus hernia, peptic ulcer, irritable bowel syndrome or esophagitis
* History of gastrointestinal surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 275 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Nausea and vomiting | Two weeks
  The primary outcome will be the comparison of incidence of nausea and vomiting in early versus delayed postoperative feeding.

SECONDARY OUTCOMES:
Change in postoperative pain | Two weeks
  Measure the change of postoperative pain between intervention and control groups using Visual Analogue Scale (VAS).
Improved hand grip strength | Two weeks
  Measure the hand grip strength using the hand grip dynamometer of the patients between intervention and control groups
Length of hospital stay | Two weeks
  Assess the length of hospital stay between intervention and control groups

IPD SHARING:
Plan to Share IPD: No
We do not have a plan to share individual participant data.

REFERENCES:
- [Result] Cordero DM, Miclau TA, Paul AV, Morshed S, Miclau T 3rd, Martin C, Shearer DW. The global burden of musculoskeletal injury in low and lower-middle income countries: A systematic literature review. OTA Int. 2020 Apr 23;3(2):e062. doi: 10.1097/OI9.0000000000000062. eCollection 2020 Jun. PMID 33937696
- [Result] Bergh C, Wennergren D, Moller M, Brisby H. Fracture incidence in adults in relation to age and gender: A study of 27,169 fractures in the Swedish Fracture Register in a well-defined catchment area. PLoS One. 2020 Dec 21;15(12):e0244291. doi: 10.1371/journal.pone.0244291. eCollection 2020. PMID 33347485
- [Result] Hemmann P, Friederich M, Korner D, Klopfer T, Bahrs C. Changing epidemiology of lower extremity fractures in adults over a 15-year period - a National Hospital Discharge Registry study. BMC Musculoskelet Disord. 2021 May 19;22(1):456. doi: 10.1186/s12891-021-04291-9. PMID 34011331
- [Result] Karkee R, Lee AH. Epidemiology of road traffic injuries in Nepal, 2001-2013: systematic review and secondary data analysis. BMJ Open. 2016 Apr 15;6(4):e010757. doi: 10.1136/bmjopen-2015-010757. PMID 27084283
- [Result] Belete Y, Belay GJ, Dugo T, Gashaw M. Assessment of Functional Limitation and Associated Factors in Adults with Following Lower Limb Fractures, Gondar, Ethiopia in 2020: Prospective Cross-Sectional Study. Orthop Res Rev. 2021 Mar 9;13:35-45. doi: 10.2147/ORR.S300459. eCollection 2021. PMID 33727867
- [Result] Sugi MT, Davidovitch R, Montero N, Nobel T, Egol KA. Treatment of lower-extremity long-bone fractures in active, nonambulatory, wheelchair-bound patients. Orthopedics. 2012 Sep;35(9):e1376-82. doi: 10.3928/01477447-20120822-25. PMID 22955405
- [Result] Hirsch KR, Wolfe RR, Ferrando AA. Pre- and Post-Surgical Nutrition for Preservation of Muscle Mass, Strength, and Functionality Following Orthopedic Surgery. Nutrients. 2021 May 15;13(5):1675. doi: 10.3390/nu13051675. PMID 34063333
- [Result] Reber E, Gomes F, Vasiloglou MF, Schuetz P, Stanga Z. Nutritional Risk Screening and Assessment. J Clin Med. 2019 Jul 20;8(7):1065. doi: 10.3390/jcm8071065. PMID 31330781
- [Result] Mu J, Wu Y, Jiang C, Cai L, Li D, Cao J. Progress in Applicability of Scoring Systems Based on Nutritional and Inflammatory Parameters for Ovarian Cancer. Front Nutr. 2022 Apr 8;9:809091. doi: 10.3389/fnut.2022.809091. eCollection 2022. PMID 35464000
- [Result] Bharadwaj S, Ginoya S, Tandon P, Gohel TD, Guirguis J, Vallabh H, Jevenn A, Hanouneh I. Malnutrition: laboratory markers vs nutritional assessment. Gastroenterol Rep (Oxf). 2016 Nov;4(4):272-280. doi: 10.1093/gastro/gow013. Epub 2016 May 11. PMID 27174435
- [Result] Chen YH, Chou CH, Su HH, Tsai YT, Chiang MH, Kuo YJ, Chen YP. Correlation between neutrophil-to-lymphocyte ratio and postoperative mortality in elderly patients with hip fracture: a meta-analysis. J Orthop Surg Res. 2021 Nov 18;16(1):681. doi: 10.1186/s13018-021-02831-6. PMID 34794459
- [Result] Nogueira PLB, Dock-Nascimento DB, de Aguilar-Nascimento JE. Extending the benefit of nutrition intervention beyond the operative setting. Curr Opin Clin Nutr Metab Care. 2022 Nov 1;25(6):388-392. doi: 10.1097/MCO.0000000000000868. Epub 2022 Aug 24. PMID 36201609
- [Result] Tong E, Chen Y, Ren Y, Zhou Y, Di C, Zhou Y, Shao S, Qiu S, Hong Y, Yang L, Tan X. Effects of preoperative carbohydrate loading on recovery after elective surgery: A systematic review and Bayesian network meta-analysis of randomized controlled trials. Front Nutr. 2022 Nov 23;9:951676. doi: 10.3389/fnut.2022.951676. eCollection 2022. PMID 36505254
- [Result] Chaudhary NK, Sunuwar DR, Sharma R, Karki M, Timilsena MN, Gurung A, Badgami S, Singh DR, Karki P, Bhandari KK, Pradhan PMS. The effect of pre-operative carbohydrate loading in femur fracture: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Aug 30;23(1):819. doi: 10.1186/s12891-022-05766-z. PMID 36042436
- [Result] Lai L, Zeng L, Yang Z, Zheng Y, Zhu Q. Current practice of postoperative fasting: results from a multicentre survey in China. BMJ Open. 2022 Jul 8;12(7):e060716. doi: 10.1136/bmjopen-2021-060716. PMID 35803620
- [Result] Fachini C, Alan CZ, Viana LV. Postoperative fasting is associated with longer ICU stay in oncologic patients undergoing elective surgery. Perioper Med (Lond). 2022 Aug 2;11(1):29. doi: 10.1186/s13741-022-00261-4. PMID 35915513
- [Result] Toms AS, Rai E. Operative fasting guidelines and postoperative feeding in paediatric anaesthesia-current concepts. Indian J Anaesth. 2019 Sep;63(9):707-712. doi: 10.4103/ija.IJA_484_19. PMID 31571683
- [Result] Rimmele T, Combourieu E, Wey PF, Boselli E, Allaouchiche B, Chassard D, Escarment J. Immediate postoperative refeeding in orthopedic surgery is safe. J Anesth. 2005;19(4):323-4. doi: 10.1007/s00540-005-0337-x. PMID 16261472
- [Result] Smith-Ryan AE, Hirsch KR, Saylor HE, Gould LM, Blue MNM. Nutritional Considerations and Strategies to Facilitate Injury Recovery and Rehabilitation. J Athl Train. 2020 Sep 1;55(9):918-930. doi: 10.4085/1062-6050-550-19. PMID 32991705
- [Result] Kim JW, Park YG, Kim JH, Jang EC, Ha YC. The Optimal Time of Postoperative Feeding After Total Hip Arthroplasty: A Prospective, Randomized, Controlled Trial. Clin Nurs Res. 2020 Jan;29(1):31-36. doi: 10.1177/1054773818791078. Epub 2018 Jul 24. PMID 30041540
- [Result] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale R, Waitzberg DL, Bischoff SC, Singer P. ESPEN guideline: Clinical nutrition in surgery. Clin Nutr. 2017 Jun;36(3):623-650. doi: 10.1016/j.clnu.2017.02.013. Epub 2017 Mar 7. PMID 28385477